CLINICAL TRIAL: NCT00460148
Title: An Open Label, Repeat Dose, Dose Escalation Study Conducted in Parkinson's Disease Patients to Characterize the Pharmacokinetics and Effect of Food on Ropinirole Prolonged Release (PR/CR) 12mg Tablets.
Brief Title: Parkinson's Disease Patient Study On Absorption, Distribution, Metabolism And Excretion Of Ropinirole
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ROP109087
Record Dates: First submitted 2007-04-11; First posted 2007-04-13 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Parkinson Disease
Keywords: ropinirole PR/CR,; pharmacokinetic,; formulation,; food effect,; SK&F101468,; PD
MeSH Terms: conditions — Parkinson Disease | interventions — ropinirole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ropinirole

SUMMARY:
This study in PD patients is designed to assess the affect food has on the absorption, distribution, metabolism and excretion of ropinirole (by dosing some patients in the fasted state and other patients following a high-fat breakfast), and to assess the difference in absorption, distribution, metabolism and excretion of ropinirole if patients are given three 4mg ropinirole tablets versus one 12mg tablet.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 30 and 85 years of age
* Body mass index of 18 to 32 kg/m2, body weight of at least 50 kg.
* Diagnosis of idiopathic Parkinson's disease
* Patients must have provided written informed consent prior to performing any study procedures
* QTc interval of < 450ms (or QTc < 480ms in patients with Bundle Branch Block).

Exclusion Criteria:

* Patients who have an abnormality on physical examination.
* Patients who have medical conditions which could present a safety concern.
* Patients who have a clinically significant abnormal laboratory value, ECG, or physical examination finding
* Positive result for Hepatitis B surface antigen, Hepatitis C antibody or Human Immunodeficiency Virus (HIV) antibody
* Positive alcohol test result and / or urine test for undeclared drugs
* Recent history of moderate to severe dizziness, syncope, or orthostatic hypotension
* Significant sleep disorder or Epworth Sleep Score (Appendix 5) > 9
* Patients with a lying/sitting diastolic blood pressure =110mmHg or =50mmHg or a systolic blood pressure =180mmHg or =90mmHg
* History of any dopaminergic treatment (other than ropinirole IR and L-dopa) within 2 weeks prior to first dose.
* Withdrawal, introduction, or change in dose of hormone replacement therapy and/or any drug known to substantially inhibit CYP1A2 or induce CYP1A2
* Patients who smoke >20 cigarettes per day and will not maintain a constant smoking habit for the duration of the study.
* Blood donation or significant blood loss less than 90 days before Day 1 of the current study.
* Definite or suspected personal history, or family history, of adverse reactions or hypersensitivity to ropinirole or to drugs with a similar chemical structure.
* Use of any investigational drug (with the exception of ropinirole PR/CR) within 30 days or 5 half lives (whichever is longer) before the start of dosing with study medication.
* Patients who have received over-the-counter (OTC) medicine within 48 h before the first dose of study drug.
* Recent history, or suspicion, of drug dependence or abuse of alcohol
* Significant concern, or likelihood, that the patient will drop out of the study prematurely, will require new or prohibited concomitant medications during the study period, or will not be compliant with study procedures.
* Women who are pregnant or breast-feeding.
* Female patient is currently either of:

  1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or any female who is surgically sterilized (via documented hysterectomy or bilateral tubal ligation).

     (For purposes of this study, postmenopausal is defined as one year without menses) OR
  2. child-bearing potential, has a negative urine/serum pregnancy test at the Screening Visit (prior to investigational product administration), and agrees to use acceptable contraception from one month prior to study Day 1 until one month after completion of the study (ie. one month after the follow-up visit). All hormonal birth control must have been administered for at least one monthly cycle prior to the Screening Visit. GSK acceptable contraception methods, when used consistently and in accordance with both the product label and the instructions of a physician, are as follows:

     * complete abstinence
     * sterilization of patient's male partner prior to female patient's entry into study
     * oral contraceptive (either combined or progestogen only)
     * any intra-uterine device with a documented failure rate of less than 1% per year
     * systemic contraception (eg. norplant system)
     * double barrier method if comprised of a spermicide with either a condom or diaphragm
* Patients with prior or current major psychosis

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-04; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Ropinirole AUC, the area under the plasma concentration-time curve over 24 hours Ropinirole maximum plasma concentration over 24 hours | 24 hours

SECONDARY OUTCOMES:
Time to attain the maximum plasma concentration Incidence of adverse events over 37 days As above, but for ropinirole metabolites | over 37 days
Vital signs, ECG and clinical laboratory data over 37 days | over 37 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Berlin, State of Berlin, Germany
- GSK Investigational Site, George, Eastern Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: ROP109087 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ROP109087 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ROP109087 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ROP109087 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: ROP109087 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: ROP109087 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: ROP109087 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register